CLINICAL TRIAL: NCT05219552
Title: Understanding the Role of Food Insecurity and Depression in Non-adherence to Option B+ Among Perinatal Kenyan Women Living With HIV: A Syndemics Approach
Brief Title: Healthy Mothers: an Intervention to Support Perinatal Women Living With HIV in Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Kenya Medical Research Institute (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: K23MH116807 (NIH); K23MH116807 (NIH)
Record Dates: First submitted 2021-12-20; First posted 2022-02-02 (Actual); Results first posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Mental Health Issue; Hiv; Breastfeeding, Exclusive
Keywords: Prevention of Mother to Child Transmission of HIV (PMTCT); exclusive breastfeeding; Women Living with HIV (WLWH); financial insecurity; food insecurity
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Breast Feeding

STUDY DESIGN:
Intervention Model Description: 20 participants recruited to the intervention group at one clinic. 20 participants simultaneously recruited to a control group at a different (but matched) clinic.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group- lactation support and unconditional cash transfers (Experimental): Women in this arm will receive personal lactation support from a professional lactation specialist at 5 time points: pregnancy and at 2-weeks, 4-weeks, 6-weeks and 3-months postpartum. Women in the intervention group will also receive monthly unconditional cash transfers of 10,000 Kenyan shillings sent directly to a a mobile phone-based money transfer service accounts associated with their personal cell phone.
  Interventions: Behavioral: personalized lactation support
- Control group- standard care (No Intervention): The women enrolled in the control arm will receive standard care at a clinic similar to, but distinct from, the intervention site.

INTERVENTIONS:
Behavioral: personalized lactation support — Our intervention design aims to address food insecurity and mental health by providing an unconditional cash transfer and lactation support across the perinatal period, when women are out of the workforce caring for their infant child. The study will include pregnant women living with HIV in Kisumu Kenya. The lactation support component will focus on milk insufficiency primarily as that has been a main concern of women we've worked with in this population, in addition to general breastfeeding support which will all be delivered in one-on-one sessions with a professional lactation consultant. The cash transfer will be delivered to women from their third trimester to 6 months postpartum. The amount of the cash transfer is based on preliminary data and consultation with key stakeholders to determine a reasonable and sufficient amount to basic living expenses during this period.
  Other Names: unconditional cash transfers
  Arms: Intervention group- lactation support and unconditional cash transfers

SUMMARY:
The investigators will recruit 40 pregnant women living with HIV divided into 2 groups (n=20 intervention group, n=20 control group). The intervention group will receive personalized lactation support and monthly unconditional cash transfers (100USD/month) from approximately 30 weeks pregnancy to approximately 6-months postpartum. The control group will receive the current standard care.

DETAILED DESCRIPTION:
In Phase One of this study, the investigators identified perceived or actual milk insufficiency, as primary barrier to exclusive breastfeeding not addressed through the current education and support being provided at the clinic. Furthermore, the investigators identified financial insecurity as a deeply-rooted threat to the health and well-being of perinatal women living with HIV and their infants across time. Based on findings from the longitudinal qualitative study, key informant interviews, focus groups with the target population and a review of the literature, the investigators developed an intervention which will be pilot tested to determine the potential impact of providing individualized support from a local lactation specialist along with monthly unconditional cash transfers (UCTs) to women living with HIV from 20-35 weeks pregnancy to 6-months postpartum.

The pilot test will be carried out among 40 pregnant women divided into 2 groups (n=20 intervention group, n=20 control group). The intervention group will receive personalized lactation support and monthly UCTs from approximately 30 weeks pregnancy to approximately 6-months postpartum. Personalized lactation support will be provided by a local, experienced lactation consultant. The support will be aimed at providing person centered care to assess for and address barriers to optimal, safe infant feeding with a focus on exclusive breastfeeding for the first 6-months postpartum. The cash transfer will be 10,000 Kenyan shillings per month. This amount is slightly less than the median amount participants in the preliminary study reported needing to meet their basic needs (13,500 Kenyan shillings) and is in line with other cash transfers completed in the area. This amount is equivalent to approximately 3.33 USD per day, or about 40% more than the World Bank's most recent poverty line estimate of 1.90 USD per person per day. This amount is lower than the estimated median monthly income for those informally employed in sectors such as retail trade or food service in Kenya (estimated at 15,000 and 30,000 Kenyan shillings monthly in rural and urban areas respectively). The investigators expect this amount will allow participants to meet many basic needs during late pregnancy and throughout the period of exclusive breastfeeding when women are largely unable to maintain gainful employment.

The control group will receive the current standard care.

The investigators will recruit women during their 20th-35th week of pregnancy and follow participants until 6-months postpartum. Survey and clinical data will be collected at baseline (20-35 weeks pregnancy), 2-weeks, 4-weeks, 6-weeks, 3-months and 6-months. Qualitative interviews will be conducted at the end of the intervention period with all 20 participants in the intervention group to evaluate the acceptability of the pilot intervention as well as to better understand how UCTs were used and the perceived impact on financial security, food security, mental health, relationships with primary partners and the ability to adhere to the prevention of mother to child transmission of HIV strategies.

ELIGIBILITY:
Inclusion Criteria:

* 20-35 weeks pregnant
* Living with HIV
* Currently prescribed antiretroviral therapy (ART)

Exclusion Criteria:

* High-risk pregnancy for reasons other than HIV status (e.g., pregnancy complications, preeclampsia, gestational diabetes, preterm labor)
* Self-reported participation in another ART adherence-related intervention study
* Unable to understand consent process
* Planning on relocating out of Nyanza province within 12 months.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-02-23 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily L Tuthill, PhD, Principal Investigator — University of California San Fransisco
Locations (2):
- Kenya (2):
  - Kisumu County Hospital, Kisumu
  - Lumumba Sub-county Hospital, Kisumu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tuthill EL, Maltby AE, Odhiambo BC, Akama E, Pellowski JA, Cohen CR, Weiser SD, Conroy AA. "I Found Out I was Pregnant, and I Started Feeling Stressed": A Longitudinal Qualitative Perspective of Mental Health Experiences Among Perinatal Women Living with HIV. AIDS Behav. 2021 Dec;25(12):4154-4168. doi: 10.1007/s10461-021-03283-z. Epub 2021 May 16. PMID 33997940
- [Background] Haushofer J, Shapiro J. THE SHORT-TERM IMPACT OF UNCONDITIONAL CASH TRANSFERS TO THE POOR: EXPERIMENTAL EVIDENCE FROM KENYA. Q J Econ. 2016 Nov;131(4):1973-2042. doi: 10.1093/qje/qjw025. Epub 2016 Jul 19. PMID 33087990
- [Result] Maltby AE, Odhiambo BC, Nyaura M, Shikari R, Tuthill EL. Feasibility, acceptability and lessons learned from an infant feeding intervention trial among women living with HIV in western Kenya. BMC Public Health. 2023 Oct 5;23(1):1930. doi: 10.1186/s12889-023-16794-2. PMID 37798696
- [Result] Tuthill EL, Maltby AE, Odhiambo BC, Hoffmann TJ, Nyaura M, Shikari R, Cohen CR, Weiser SD. "It has changed my life": unconditional cash transfers and personalized infant feeding support- a feasibility intervention trial among women living with HIV in western Kenya. Int Breastfeed J. 2023 Nov 27;18(1):64. doi: 10.1186/s13006-023-00600-1. PMID 38012644

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Group- Lactation Support and Unconditional Cash Transfers | Control Group- Standard Care
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The analysis population is the same as the assignment in Participant Flow. Baseline data for participants is reported under outcome meassures.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group- Lactation Support and Unconditional Cash Transfers | Control Group- Standard Care | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 27.95 [20 to 43] | 28.5 [19 to 38] | 28 [19 to 43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 20 | 40
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Kenya | 20 | 20 | 40
Patient Health Questionnaire-9 [Median (Inter-Quartile Range); unit: score on a scale] — Patient Health Questionnaire-9: scoring ranges from 0-27 with higher scores indicating greater depressive symptoms.
  score on a scale | 8.5 [6.0 to 9.2] | 6.5 [5.0 to 9.8] | 8 [5.0 to 9.5]

OUTCOME MEASURES:

1. Primary Outcome: Maternal Mental Health
Description: Patient Health Questionnaire-9: scoring ranges from 0-27 with higher scores indicating greater depressive symptoms.
Time Frame: baseline (20-35 weeks pregnant), 6-weeks postpartum and 6-months postpartum
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention Group- Lactation Support and Unconditional Cash Transfers | Control Group- Standard Care
Number analyzed (Participants) | 20 | 20
score on a scale
  Baseline | 8.5 [6.0 to 9.2] | 6.5 [5 to 9.8]
  6 weeks postpartum | 3.0 [2 to 6.2] | 3.0 [.8 to 5]
  6 months postpartum | 3.0 [1 to 5.2] | 5 [1 to 8]

2. Primary Outcome: Number of Participants Who Reported Feeding Breastmilk Only
Description: Breast feeding behavior questionnaires where participants were asked, "What are you currently feeding your baby". The count of participants is the number of participants who selected, "breastmilk only".
Time Frame: 2 weeks, 4 weeks, 6 weeks, and 12 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group- Lactation Support and Unconditional Cash Transfers | Control Group- Standard Care
Number analyzed (Participants) | 20 | 20
Participants
  2 weeks | 19 | 16
  4 weeks | 19 | 19
  6 weeks | 20 | 19
  12 weeks | 20 | 17

3. Primary Outcome: Number of Participants Who Acknowledge Missing One or More HIV Infant Medications
Description: Questionnaire on adherence to infant HIV prophylaxis- participant count is the number of participants who acknowledged missing one more more dose of their infant's HIV medications (collected at 6 weeks and 6 months).
Time Frame: 6-weeks postpartum and 6-months postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group- Lactation Support and Unconditional Cash Transfers | Control Group- Standard Care
Number analyzed (Participants) | 20 | 20
Participants
  6 weeks | 0 | 0
  6 months | 2 | 2

4. Primary Outcome: Maternal Adherence to HIV Medications
Description: Questionnaire on Maternal Adherence to HIV medications- the reported data comes from a visual analog scale where participants were instructed, "Please point or mark at the point showing how much of your ARVs you have taken in the past 30 days."
Time Frame: baseline (20-35 weeks pregnant), 6-weeks postpartum and 6-months postpartum
Measure: Mean (Standard Deviation); unit: percentage of HIV medications taken
Arm/Group | Intervention Group- Lactation Support and Unconditional Cash Transfers | Control Group- Standard Care
Number analyzed (Participants) | 20 | 20
percentage of HIV medications taken
  Baseline | 98.95 (3.94) | 98.05 (6.95)
  6 weeks | 97.7 (10.03) | 99.75 (1.09)
  6 months | 99.8 (0.6) | 99.85 (0.48)

5. Primary Outcome: Food Security
Description: Household Food Insecurity Access scale: scoring ranges from 0-27 with higher scores indicating greater food insecurity.
Time Frame: baseline (20-35 weeks pregnant), 6-weeks postpartum and 6-months postpartum
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Intervention Group- Lactation Support and Unconditional Cash Transfers | Control Group- Standard Care
Number analyzed (Participants) | 20 | 20
units on a scale
  Baseline | 11.5 [9 to 16.2] | 12 [7 to 15]
  6 weeks postpartum | 1 [0 to 7] | 9.5 [5.8 to 12.5]
  6 months postpartum | 2 [0 to 3.5] | 9 [6 to 11.5]

6. Primary Outcome: Financial Security
Description: These data were collected qualitatively using in depth exit interviews with intervention only participants to better understand how the cash transfer was used, what changes resulted in their lives related to increased financial security due to the cash transfer.
Time Frame: 7 months
Population: Financial security was assessed qualitatively using in depth interviews at an exit interview after intervention completion
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group- Lactation Support and Unconditional Cash Transfers | Control Group- Standard Care
Number analyzed (Participants) | 20 | 0
Participants
  Exit Interview Improved Financial Security related to cash transfer intervention | 20 |
  Exit Interview No improvements to financial security related to cash transfer intervention | 0 |

7. Secondary Outcome: Relationships Status
Description: Couples satisfaction Index: scoring ranges from 0-81 with higher scores indicating greater relationship satisfaction.
Time Frame: baseline (20-35 weeks pregnant), 6-weeks postpartum and 6-months postpartum
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group- Lactation Support and Unconditional Cash Transfers | Control Group- Standard Care
Number analyzed (Participants) | 20 | 20
score on a scale
  Baseline | 41.3 (11.6) | 44.5 (22.2)
  6 weeks | 44.4 (14.8) | 53.3 (11.6)
  6 months | 43.1 (15.5) | 50.3 (10.8)

8. Secondary Outcome: Women's Empowerment
Description: Select questions from the Demographic Health Survey-"Who usually decides how the money you earn will be used: mainly you, mainly your husband/partner, or you and your husband/partner jointly?" and a series of questions asking if the participants current partner has been verbally, physically and/or sexually abusive over the preceding 12 months.
Time Frame: baseline (20-35 weeks pregnant), 6-weeks postpartum and 6-months postpartum
Population: Some participants chose the option "not applicable" for the decision making question since they were not "earning" any money. Also, data are missing from several participants on the questions about experience of abuse- see # of participants analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group- Lactation Support and Unconditional Cash Transfers | Control Group- Standard Care
Number analyzed (Participants) | 20 | 20
Participants
  Baseline -mainly participant decides | 9 | 11
  Baseline- mainly husband/ partner decides | 1 | 2
  Baseline - decides jointly | 0 | 7
  Baseline- other | 10 | 0
  6 weeks -mainly participant decides | 6 | 11
  6 weeks- mainly husband/ partner decides | 0 | 1
  6 weeks - decides jointly | 3 | 8
  6 weeks-other | 11 | 0
  6 months -mainly participant decides | 7 | 14
  6 months -mainly husband/ partner decides | 0 | 2
  6 months -decides jointly | 6 | 4
  6 months- other | 7 | 0
  Baseline- has experienced abuse by husband/partner | 13 | 14
  6 weeks- has experienced abuse by husband/partner: number analyzed (Participants) | 20 | 19
  6 weeks- has experienced abuse by husband/partner | 10 | 10
  6 months- has experienced abuse by husband/partner: number analyzed (Participants) | 19 | 18
  6 months- has experienced abuse by husband/partner | 10 | 9

9. Secondary Outcome: HIV-related Stigma
Description: 12-item HIV stigma scale: scoring ranges from 12-48 higher scores reflect a higher level of perceived HIV-related stigma.
Time Frame: baseline (20-35 weeks pregnant), 6-weeks postpartum and 6-months postpartum
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group- Lactation Support and Unconditional Cash Transfers | Control Group- Standard Care
Number analyzed (Participants) | 20 | 20
score on a scale
  Baseline | 25.6 (6.3) | 30.4 (7.1)
  6 weeks | 25.9 (3.9) | 27.1 (4.6)
  6 months | 26.8 (4.1) | 28.4 (4.7)

10. Secondary Outcome: Social Support
Description: Duke-University of North Carolina Functional Social Support Questionnaire: scoring ranges from 8-40 with higher values indicating greater social support
Time Frame: 6-weeks postpartum and 6-months postpartum
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention Group- Lactation Support and Unconditional Cash Transfers | Control Group- Standard Care
Number analyzed (Participants) | 20 | 20
score on a scale
  6 weeks | 24.5 [20.2 to 31.5] | 33.0 [27.8 to 37.0]
  6 month | 30.5 [22.0 to 34.0] | 31.0 [27.8 to 35.5]

ADVERSE EVENTS:
Time Frame: Between 8-11months depending on when a participant was recruited (recruitment was from 20-35weeks pregnant) and the time of their infants birth. Therefore, participants were assessed over a period from 8-11 months.
Groups:
- Intervention Group- Lactation Support and Unconditional Cash Transfers: Women in this arm will receive personal lactation support from a professional lactation specialist at 5 time points: pregnancy and at 2-weeks, 4-weeks, 6-weeks and 3-months postpartum. Women in the intervention group will also receive monthly unconditional cash transfers of 10,000 Kenyan shillings sent directly to a a mobile phone-based money transfer service accounts associated with their personal cell phone.
  personalized lactation support: Our intervention design aims to address food insecurity and mental health by providing an unconditional cash transfer and lactation support across the perinatal period, when women are out of the workforce caring for their infant child. The study will include pregnant women living with HIV in Kisumu Kenya. The lactation support component will focus on milk insufficiency primarily as that has been a main concern of women we've worked with in this population, in addition to general breastfeeding support which will all be delivered in one-on-one sessions with a professional lactation consultant. The cash transfer will be delivered to women from their third trimester to 6 months postpartum. The amount of the cash transfer is based on preliminary data and consultation with key stakeholders to determine a reasonable and sufficient amount to basic living expenses during this period.
  0 Adverse Events
- Control Group- Standard Care: The women enrolled in the control arm will receive standard care at a clinic similar to, but distinct from, the intervention site.
  0 Adverse Events
Arm/Group | Intervention Group- Lactation Support and Unconditional Cash Transfers | Control Group- Standard Care
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-09-14): https://cdn.clinicaltrials.gov/large-docs/52/NCT05219552/Prot_001.pdf
  • Informed Consent Form (2021-10-08): https://cdn.clinicaltrials.gov/large-docs/52/NCT05219552/ICF_002.pdf